CLINICAL TRIAL: NCT07102589
Title: Predictive Value of the Shuttle Walking Test for Postoperative Dyspnea in Chronic Respiratory Disease Patients Undergoing Lung Resection: A Prospective Observational Study
Brief Title: SWEEP: Shuttle Walking Test for Exercise Evaluation in Pulmonary Resection
Acronym: SWEEP
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SWEEP-PRO-SNUBH-01; B-2506-980-301 (Registry Identifier: SNUBH IRB (Seoul National University Bundang Hospital Institutional Review Board))
Record Dates: First submitted 2025-07-30; First posted 2025-08-04 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-06

CONDITIONS: COPD; ILD; Bronchiectasis; Lung Cancer NOS; Dyspnea During Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study that evaluates whether the Shuttle Walking Test (SWT) can predict postoperative symptoms, particularly dyspnea, in patients with chronic respiratory diseases undergoing lung resection.

Currently, tools such as DLCO or cardiopulmonary exercise testing (CPET) are used to assess surgical risk and exercise capacity before lung surgery. However, these tests are not always accessible due to equipment limitations or long waiting times. The SWT is a simpler, safer, and more cost-effective alternative that has been recently recognized as a new medical technology in Korea for evaluating exercise capacity.

In this study, patients with chronic lung diseases (such as COPD, ILD, or bronchiectasis) who are scheduled to undergo lung resection will perform the SWT before surgery. Their symptoms and quality of life will be assessed through questionnaires before and three months after the surgery. The goal is to determine whether SWT results can help predict postoperative dyspnea and provide useful information for preoperative risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 40 years
* Scheduled for surgical lung resection (e.g., for lung cancer or benign tumor)
* Diagnosis of chronic respiratory disease (COPD, ILD, or bronchiectasis)
* Able to perform Shuttle Walking Test (ISWT + ESWT) before surgery
* Able to complete pre- and postoperative symptom questionnaires (dyspnea, EQ-5D)

Exclusion Criteria:

* - Illiteracy or inability to read study materials
* Inability to communicate in Korean
* Decline or withdraw consent
* Severe lower limb disability interfering with walking (e.g., fracture, paralysis)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 19 years or older with chronic respiratory diseases (such as COPD, ILD, or bronchiectasis) who are scheduled to undergo surgical lung resection at Seoul National University Bundang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dyspnea Score From Baseline to 3 Months After Lung Resection | From baseline (preoperative) to 3 months postoperatively
  Dyspnea will be assessed using a validated scale (e.g., POSPNEA or MRC). The difference in scores between preoperative baseline and 3 months after surgery will be analyzed.
Predictive Value of Shuttle Walking Test for Postoperative Dyspnea | Preoperative to 3 months postoperative
  The correlation between preoperative SWT results (ISWT distance, endurance time) and postoperative dyspnea score at 3 months will be evaluated using regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Not Required For This Country, South Korea